CLINICAL TRIAL: NCT06717997
Title: The Third-trimester Placental Thickness and Pregnancy Outcomes in Placenta Previa Women
Brief Title: The Placental Thickness and Pregnancy Outcomes in Placenta Previa Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Assistant Professor, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PAS-US
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal placental thickness women (Other)
  Interventions: Other: ultrasound
- High placental thickness women (Other)
  Interventions: Other: ultrasound

INTERVENTIONS:
Other: ultrasound — The placenta thickness will be performed on transabdominal images obtained in a longitudinal plane. Three measurements will be performed at the thickest portion of the placenta. The average of these three measurements was used for statistical analysis. The cohorts will be classified into 1) thick placenta (>4 cm) and average placenta (2-4 cm).

SUMMARY:
Placenta previa is the placenta overlying the cervical os. Placenta previa is about 1 in 200 pregnancies. The risk factors are the increasing rate of cesarean section and previous uterine surgery. Placenta previa is associated with many adverse complications; the most serious one is related to maternal hemorrhage. The diagnosis of placenta previa is done by trans-abdominal and trans-vaginal ultrasonography, which can document the placental edge's relationship to the internal os. Placenta accreta spectrum disorder is defined when trophoblastic invades the myometrium. The Placenta accreta spectrum can be categorized as: placenta accreta, placenta increta, and placenta percreta.

The clinical utility of placental thickness is an area of ongoing research in placenta previa. Prior studies have demonstrated an association between mid-trimester placental thickness and placenta accreta spectrum. Despite the presence of many studies in characterizing placental thickness, most studies have focused primarily on the placental accreta spectrum lacking information about other fetal and maternal complications. Symptomatic (bleeding) placenta previa is associated with increased maternal and neonatal morbidity and mortality. In addition; the mechanism that involves bleeding is unclear. It is usually related to uterine contractions, cervical effacement, and dilation leading to separation of the placenta from the underlying decidua.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women from 32-34 weeks.
2. Pregnant women with singleton pregnancy.
3. Women with placenta previa.
4. Placenta previa with minimal vaginal bleeding or haven't any vaginal bleeding.
5. Women without any medical disorders.
6. Women should be living in a nearby area to make follow-up and early transportation is reasonably possible.

Exclusion Criteria:

1. Women with severe bleeding necessitate immediate delivery.
2. Women with confirmed fetal malformation.
3. If associated with abruptio placentae.
4. Women who will refuse to participate.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
number of women with placenta accreta | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided